CLINICAL TRIAL: NCT05495789
Title: The Effect of Virtual Reality and Music Application on Non-Stress Test Parameters, Anxiety and Satisfaction During Non-Stress Test in High-Risk Pregnants
Brief Title: The Effect of Virtual Reality and Music in High-Risk Pregnants on Non-Stress Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NESLİHAN YILMAZ SEZER (Other)
Responsible Party: Sponsor-Investigator, NESLİHAN YILMAZ SEZER, Faculty of Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12/125
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: High Risk Pregnancy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): In addition to the routine procedure, virtual reality glasses will be applied to the high-risk pregnant in the virtual reality group of the research. Virtual reality glasses is a device that works on compatible smart mobile phones. After the NST device is connected and, the high-risk pregnant included in the experimental group will be made to watch a video lasting an average of 40 minutes with virtual reality glasses until the procedure is completed.
  Interventions: Other: Virtual Reality
- Music Group (Experimental): In addition to the routine procedure, the high-risk pregnant women in the music group of the research will listen to the relaxing music used in the virtual reality application with headphones.
  Interventions: Other: Music
- Control Group (No Intervention): The high-risk pregnants in the control group of the study will not be subjected to any treatment other than the routine procedure.

INTERVENTIONS:
Other: Virtual Reality — A relaxing video will be watched with virtual reality glasses.
  Arms: Virtual Reality Group
Other: Music — Relaxing music will be played by wearing headphones.
  Arms: Music Group

SUMMARY:
Aim: The aim of this study is to determine the effects of virtual reality and listening to music during the NST procedure on NST parameters, anxiety and satisfaction in high-risk pregnant.

Hypotheses H01 In the NST process, there is no difference between the NST parameters of the virtual reality group and the NST parameters of the control group.

H02 In the NST procedure, there was no difference between the anxiety score of the virtual reality group and the anxiety score of the control group.

H03 There is no difference between the satisfaction score of the group in which virtual reality was applied in the NST procedure and the satisfaction score of the control group.

H04 In the NST process, there is no difference between the NST parameters of the group to which the virtual reality is applied and the NST parameters of the musical group.

H05 In the NST procedure, there was no difference between the anxiety score of the group in which virtual reality was applied and the anxiety score of the music group.

H06 In the NST process, there is no difference between the satisfaction score of the group to which the virtual reality was applied and the satisfaction score of the music group.

H07 In NST operation, there is no difference between the NST parameters of the music group and the NST parameters of the control group.

H08 In the NST procedure, there was no difference between the anxiety score of the music group and the anxiety score of the control group.

H09 There is no difference between the satisfaction score of the music group and the satisfaction score of the control group in the NST procedure.

DETAILED DESCRIPTION:
The study will be carried out in three different groups. The practice will start with meeting the high-risk pregnant who apply to the NST. After the women are evaluated in terms of eligibility criteria for the research, the high-risk pregnant who are eligible will be informed about the research and written informed consent will be obtained from the high-risk pregnant who accept. The random distribution of high-risk pregnant to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Virtual Reality Group In addition to the routine procedure, virtual reality glasses will be applied to the high-risk pregnant in the virtual reality group of the research. Virtual reality glasses is a device that works on compatible smart mobile phones. After the NST device is connected and, the high-risk pregnant included in the experimental group will be made to watch a video lasting an average of 40 minutes with virtual reality glasses until the procedure is completed.

Music Group In addition to the routine procedure, the high-risk pregnant women in the music group of the research will listen to the relaxing music used in the virtual reality application with headphones.

Control Group The high-risk pregnants in the control group of the study will not be subjected to any treatment other than the routine procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being at the 32nd and above gestational week
* Pregnant women with a single fetus
* Have eaten at least two hours before the NST procedure
* No cardiovascular disease diagnosed in the fetus,
* The participants ate at least 2 h before the NST, urinated immediately before the NST and did not smoke or drink alcohol for at least 2 h before the NST.
* Those diagnosed with high-risk pregnancy by a physician (pregnancy-induced hypertension, preeclampsia, eclampsia, gestational diabetes, premature rupture of membranes, pregnancy large or small for gestational age, intrauterine growth retardation, polihydramnios, oligohydramnios, premature birth threat, maternal age 35 age and above, maternal body mass index over 30 (obesity)
* Not having vision and hearing problems

Exclusion Criteria:

* Pregnant women with major medical (cardiac, renal or neurological diseases) or mental illnesses (psychosis, neurosis, addictions, etc.)
* healty pregnant women
* multiple pregnancy
* having a fetus with anomaly,
* Pregnant women with fetal distress and for whom emergency intervention is considered by the physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | immediately before the NST procedure and immediately after the NST procedure
  STAI-S consist of 20 items with four points Likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
the degree of satisfaction | immediately after the NST procedure
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfied and a score of 0 pointed to no satisfied.
Non-Stress Test Parameters/ basal fetal heart rate | immediately after the NST procedure
  It is the average fetal heart rate sustained over a 10-minute period and 120-160 beats/minute is normal.
Non-Stress Test Parameters: number of accelerations | immediately after the NST procedure
  Acceleration an increase in fetal heart rate.
Non-Stress Test Parameters/ number of decelerations | immediately after the NST procedure
  Deceleration is the slowing of fetal heart rate seen on the monitor during contractions.
Non-Stress Test Parameters/ reactive nst | immediately after the NST procedure
  Reactive NST; It is a normal result showing that accelerations occur at least twice within a maximum of 20 minutes, are at least 15 beats/min more than the basal level and continue for 15 seconds.
Non-Stress Test Parameters / Test time (minutes) for reactive NST | immediately after the NST procedure
  Time until reactive NST result is obtained.
Non-Stress Test Parameters / Non-reaktif NST | immediately after the NST procedure
  Non-reactive NST; An abnormal result showing that less than two of the accelerations that are at least 15 beats/min above baseline occur in a 40 min time frame.

CONTACTS AND LOCATIONS:
Overall Officials: AYKAN YÜCEL, Prof.Dr., Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Neslihan Yılmaz Sezer, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No